CLINICAL TRIAL: NCT00092326
Title: A Randomized, Double-Blind, Placebo- and Active-Comparator-Controlled Study to Evaluate the Efficacy of Rofecoxib and a Dosing Regimen of Oxycodone With Acetaminophen Over 24 Hours in Patients With Postoperative Dental Pain
Brief Title: A Study of Two Approved Drugs in the Treatment of Postoperative Dental Pain (0966-183)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-183; 2004_068
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Pain
Keywords: dental surgery; molar removal
MeSH Terms: conditions — Pain, Postoperative | interventions — rofecoxib; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0966, rofecoxib
Drug: Comparator: oxycodone with acetaminophen, placebo

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two approved drugs in the treatment of pain following dental surgery.

DETAILED DESCRIPTION:
The duration of treatment is 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Impaction of a molar tooth requiring removal

Exclusion Criteria:

* Any known allergy to the study drugs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2002-06; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Post-op dental pain over 6 hours as measured by pain intensity/relief scores, patient global assessment, and time to perceptible/meaningful pain relief.

SECONDARY OUTCOMES:
Time to onset of analgesic effect, peak analgesic effect, and/or duration of analgesic effect over 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Desjardins PJ, Black PM, Daniels SE, Bird SR, Petruschke RA, Chang DJ, Smugar SS, Tershakovec AM. A double-blind randomized controlled trial of rofecoxib and multidose oxycodone/acetaminophen in dental impaction pain. J Oral Maxillofac Surg. 2007 Aug;65(8):1624-32. doi: 10.1016/j.joms.2006.06.268. No abstract available. PMID 17656293